CLINICAL TRIAL: NCT00216372
Title: Phase III, Multicentre, Randomised, Double-blind, Comparative Study to Assess the Efficacy and Safety of Lanreotide 30 mg Versus Placebo as a Palliative Treatment of Clinical Symptoms Associated With Intestinal Obstruction Due to Peritoneal Carcinomatosis in Inoperable Patients.
Brief Title: Efficacy and Safety of Lanreotide Microparticles as Palliative Treatment in Peritoneal Carcinomatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-54-52030-156 (408); 2005-002349-38 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Intestinal Obstruction; Carcinoma; Peritoneal Neoplasms
Keywords: carcinomatosis
MeSH Terms: conditions — Intestinal Obstruction; Carcinoma; Peritoneal Neoplasms | interventions — lanreotide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Lanreotide (microparticle formulation)
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lanreotide (microparticle formulation) — A single 30 mg intra-muscular injection on day 0. The duration of the blinded phase is 10 days. Patients may enter the open phase where they receive 30 mg intra-muscular injections, every 10 days until investigator/or patient decide to stop treatment.
  Arms: 1
Other: Placebo — A single intra-muscular injection on day 0.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether lanreotide 30mg microparticles are effective in the relief of clinical symptoms due to small bowel obstruction in inoperable patients with peritoneal carcinomatosis.

ELIGIBILITY:
Inclusion Criteria:

* digestive obstruction located in the upper part of the gastro-intestinal tract
* digestive obstruction of malignant origin
* peritoneal carcinomatosis confirmed by a CT Scan
* at least two vomiting episodes per day or a presence of a nasogastric suction tube
* inoperable patients

Exclusion Criteria:

* specific anticancer therapy within the previous 15 days
* signs of bowel perforation
* somatostatin or any analogue as treatment of the bowel obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2003-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Percentage of responder patients (patient with 1 or less vomiting episode per day during at least 3 consecutive days or in whom nasogastric tube (NGT) has been removed during at least three consecutive days without vomiting recurrence) | On day 7 (plus 1 day at the latest) after the first injection

SECONDARY OUTCOMES:
Number of daily vomiting episodes or measurement of the daily drainage by NGT | Daily for the duration of the study
Number of days with no vomiting episodes | For the duration of the study
Number of daily nausea episodes | Daily for the duration of the study
Intensity of abdominal pain | Daily for the duration of the study
Well-being | Daily for the duration of the study
Symptom relief duration | Between the first day of clinical response and the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (53):
- Belgium (4):
  - Clinique Universitaire St. LUC, Brussels
  - Institut Jules Bordet, Brussels
  - Clinique Notre-Dame, Hermalle-sous-Huy
  - Centre Hospitalier de Jolimont-Lobbes, La Louvière
- France (48):
  - Hôpital Nord, Amiens
  - Clinique de l'Anjou, Angers
  - Hôtel-Dieu, Angers
  - CH Victor Dupouy, Argenteuil
  - Hôpital Saint André, Bordeaux
  - Hôpital de la Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Hôpital Nord, Cébazat
  - Clinique de l'Amandier, Châtenay-Malabry
  - Hôpital Hôtel-Dieu, Clermont-Ferrand
  - Hôpital Beaujon, Clichy
  - Hôpital Pasteur, Colmar
  - Centre Hospitalier de Compiègne, Compiègne
  - Hôpital Henri Mondor, Créteil
  - Centre Hospitalier Victor Jousselin, Dreux
  - Clinique Sainte Marguerite, Hyères
  - Centre Hospitalier Départemental, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - Hôpital Notre-Dame du Perpétuel Secours, Levallois-Perret
  - CHU Dupuytren, Limoges
  - Hôpital Site de Lorient, Lorient
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital de l'Archet 2, Nice
  - Hôpital de la Source, Orléans
  - Centre de Radiothérapie et Oncologie Médicale, Osny
  - Hôpital du Val de Grâce, Paris
  - Institue Curie, Paris
  - Hôpital des Diaconesses, Paris
  - Hôpital Saint Antoine, Paris
  - Hôtel Dieu, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier de Roanne, Roanne
  - CAC Becquerel, Rouen
  - Hôpital Charles Nicolle, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Clinique Guillaume de Varye, Saint-Doulchard
  - Institut de Cancérologie de la Loire, Saint-Etienne
  - Centre Hospitalier Gaston Ramon, Sens
  - Hôpital Civil, Strasbourg
  - Hôpital Hautepierre, Strasbourg
  - C.H.R. de Metz-Thionville, Thionville
  - Hôpital de Rangueil, Toulouse
  - Hôpital Joseph Ducuing, Toulouse
  - Institut Gustave Roussy, Villejuif
- Academisch Medisch Centrum, Amsterdam, Netherlands

REFERENCES:
- [Derived] Mariani P, Blumberg J, Landau A, Lebrun-Jezekova D, Botton E, Beatrix O, Mayeur D, Herve R, Maisonobe P, Chauvenet L. Symptomatic treatment with lanreotide microparticles in inoperable bowel obstruction resulting from peritoneal carcinomatosis: a randomized, double-blind, placebo-controlled phase III study. J Clin Oncol. 2012 Dec 10;30(35):4337-43. doi: 10.1200/JCO.2011.40.5712. Epub 2012 Oct 29. PMID 23109694